CLINICAL TRIAL: NCT06202716
Title: Cadonilimab Plus CapeOX as First-Line Treatment for Advanced GC/GEJC With High Tumor Microenvironment Score (TMEscore).
Brief Title: Cadonilimab Plus CapeOX as First-Line Treatment for Advanced GC/GEJC With High TMEscore
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-531
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: Cadonilimab; CapeOX; First-line treatment; GC/GEJC; TMEscore
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab plus CapeOX chemotherapy (Experimental): Efficacy of cadonilimab plus CapeOX as first-line treatment in advanced GC/GEJC with high TMEscore.
  Interventions: Drug: Cadonilimab plus CapeOX chemotherapy

INTERVENTIONS:
Drug: Cadonilimab plus CapeOX chemotherapy — Cadonilimab plus oxaliplatin/capecitabine (CapeOX) chemotherapy as first-line treatment in patients with advanced gastric cancer or gastro-esophageal junction adenocarcinoma: Cadonilimab 10mg/kg, iv, q3w + oxaliplatin 130mg/m2, vd, d1 + capecitabine 1000mg/m2, po, bid, d1-d4, q3w (3 weeks as a cycle, a maximum of 8 cycles of treatment). Then the maintenance treatment phase with tislelizumab + lenvatinib is entered, and the specific dosage is the same as the treatment period.

SUMMARY:
This is a single-arm, open-label, multi-center clinical study to evaluate the efficacy and safety of PD-1/CTLA-4 bispecific cadonilimab in combination with oxaliplatin/capecitabine (CapeOX) in the first-line treatment of advanced gastric cancer or gastro-esophageal junction adenocarcinoma with a high tumor microenvironment score (TMEscore). The study plans to enroll 50 patients to receive cadonilimab 100mg/kg, iv, q3w + CapeOX (oxaliplatin 130mg/m2, vd, d1 + capecitabine 1000mg/m2, po, bid, D1-14, q3w, with 3 weeks as a cycle and a maximum of 8 cycles of treatment. Then the maintenance treatment phase with cadonilimab ± capecitabine is entered, and the specific dosage is the same as the treatment period. Effectiveness is assessed every 9 weeks (±7 days) using RECISIT 1.1 until disease recurrence, metastasis, death, or loss of follow-up. The primary endpoint of this study was PFS, and secondary endpoints were OS, ORR, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study, sign the informed consent form, and have good compliance;
2. Age≥ 18 years old, gender is not limited;
3. Histologically confirmed locally advanced unresectable or advanced metastatic adenocarcinoma of the stomach and gastroesophageal junction;
4. The tumor tissue was tested by the tumor microenvironment in the laboratory of the Department of Oncology, Nanfang Hospital, Southern Medical University, and was defined as a high tumor microenvironment score (TMEscore).
5. Her2 negative or ambiguous;
6. No prior systemic first-line therapy;
7. Subjects who have received prior adjuvant chemotherapy or neoadjuvant chemotherapy with curative intent or definitive chemo-radiotherapy for advanced disease are eligible if progression occurs >6 months after the previous treatment;
8. ECOG physical condition 0 or 1 point;
9. Expected survival ≥ 3 months;
10. Blood tests (without transfusion within 14 days) 1) Absolute neutrophil ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥90g/L); 2) Liver function tests (aspartate aminotransferase and glutamate aminotransferase ≤3× ULN, bilirubin ≤1.5×ULN; in case of liver metastases, AST and ALT ≤5×ULN); 3) renal function (serum creatinine ≤ 1.5×ULN, or creatinine clearance (CCr) ≥60ml/min);
11. Men and women of childbearing age must use effective contraception

Exclusion Criteria:

1. Squamous cell carcinoma, undifferentiated or other non-adenocarcinoma histologic type of gastric cancer or gastro-esophageal tumor;
2. Subjects with known contraindications to cadonilimab, CapeOX (see package inserts for cadonilimab, oxaliplatin, and capecitabine);
3. Known history of severe intolerance to cadonilimab, oxaliplatin, or capecitabine (i.e., grade 4 toxicity of one of the agents; grade 3-4 toxicity of other concomitant agents is not excluded);
4. Known history of hypersensitivity or hypersensitivity to cadonilimab, oxaliplatin, other platinum compounds, or fluorouracil;
5. Known brain or meningeal metastases:
6. Radiotherapy or any anti-tumor therapy (chemotherapy, targeted therapy, immunotherapy, radio-frequency ablation, traditional Chinese medicine with anti-tumor indications, immunomodulators or tumor embolization, etc.) within 4 weeks prior to the first dose of study treatment;
7. Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies, or any other antibody or drug therapy against T cell co-stimulation or checkpoint pathways;
8. Patients have had other malignancies within the past 5 years or at the same time (except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
9. There are obvious clinical bleeding symptoms or obvious bleeding tendency, hemoptysis, etc. within 3 months before treatment. or venous/venous thrombotic event treatment within the preceding 6 months, such as cerebrovascular accident (including transient ischemic attack, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; or requiring long-term anticoagulation with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin≥ 300 mg/day or clopidogrel ≥75 mg/day);
10. Active heart disease, including myocardial infarction, severe/unstable angina, 6 months prior to treatment. Echocardiography of left ventricular ejection fraction <50%;
11. Known history of primary or secondary immunodeficiency virus infection
12. Concomitant active or uncontrolled severe infection
13. Any other disease, clinically significant metabolic abnormality, physical examination abnormality, or laboratory abnormality that, in the judgment of the investigator, has reason to suspect that the patient has a certain disease or state that is not suitable for the use of the study drug;
14. Any condition that, in the opinion of the investigator, may put subjects treated with study drug at risk, interfere with the study drug, subject safety assessment, or interpretation of results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 3 years
  Defined as the time between the onset of PD or death when a patient first receives the study drug, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Defined as the time between the patient's first receipt of the study drug to death.
Objective Response Rate (ORR) | 3 years
  Defined as the proportion of patients who achieved complete response (CR) or partial response (PR).
Safety | 3 years
  The occurrence of various AEs, including SAEs, will be monitored based on changes in various indicators such as vital signs, physical examination, 12-lead electrocardiogram (ECG), laboratory tests, etc. AEs will be graded for severity according to NCI CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No